CLINICAL TRIAL: NCT01981707
Title: F-choline PET in Early Response Assessment for Castration Resistant Prostatic Cancer Treated by Abiraterone Acetate or Enzalutamide
Brief Title: F-choline PET in Early Response Assessment for Castration Resistant Prostatic Cancer
Acronym: PRECHOL
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: enrollment default
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2013-003058-25
Record Dates: First submitted 2013-08-01; First posted 2013-11-11 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-04

CONDITIONS: Castration-resistant Prostate Cancer
Keywords: castration-resistant prostate cancer; abiraterone acetate; enzalutamide; choline pet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- F-Choline PET (Experimental): The F-Choline-PET will be performed before and at 6 weeks of the beginning of treatment by abiraterone acetate or enzalutamide.
  Interventions: Device: F-Choline-PET

INTERVENTIONS:
Device: F-Choline-PET

SUMMARY:
Until today no current diagnostic tool exists to identify an early objective response when patients with castration-resistant prostate cancer were treated by abiraterone acetate or enzalutamide. According to the Prostate Cancer Working Group, the investigators have to wait 12 weeks before the first evaluation. To know soon that the treatment is effective will be decisive for the oncologist, even more in palliative situation where second effects can't be imposed to patients.

In post-docetaxel, the F-choline PET-CT could be used to assess the response of this new therapy. Moreover, the investigators suppose that we can assess an early stage if there is an objective therapeutic response, at 6 weeks of treatment, in order to avoid unnecessarily and expansive treatment.

The aim of this study is to assess if it is possible to determine early (6 weeks of treatment)if a F-choline PET-CT could predict the response to abiraterone acetate or enzalutamide in post-docetaxel.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Eastern Cooperative Oncology Group (ECOG)performance status score of 2 or less
* Histologically or cytologically confirmed adenocarcinoma prostate cancer without neuroendocrine component (component with minority neuroendocrine) or small cell, or neuroendocrine cells or small minority component prostate who underwent surgical or medical castration
* Disease progression during or after a docetaxel-based chemotherapy
* serum testosterone level of 50 ng per deciliter or less (≤2.0 nmol per liter)
* Biologic criteria :
* platelets ≥ 100 000/μl,
* Creatinine <1.5 x upper limit or creatinine clearance ≥ 60 ml / min,
* Serum potassium ≥ 3.5 mmol / l,
* Bilirubin <1.5 x upper limit of normal (ULN)
* hemoglobin ≥ 9.0 g / dl without any transfusion.

Exclusion Criteria:

* abnormal aminotransferase levels (levels of aspartate aminotransferase or alanine aminotransferase that were ≥2.5 times the upper level of the normal range; patients with known liver metastasis who had levels of aspartate aminotransferase or alanine aminotransferase that were ≤5 times the upper level of the normal range were eligible to participate
* previous therapy with ketoconazole
* serious coexisting nonmalignant disease :
* active or symptomatic viral hepatitis or chronic liver disease,
* uncontrolled hypertension,
* a history of pituitary or adrenal dysfunction,
* clinically significant heart disease

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-12; Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of 6 weeks PET-CT performed on the response after 12 weeks of abiraterone acetate treatment or enzalutamide | 12 weeks
  A centralized review will be carried out by 2 independent reviewers. The gold-standard to evaluate tumoral response to abiraterone acetate or enzalutamide will be the pain, the Prostate Specific Antigen rate, and imagery at 3 months according to prostate cancer working group.

SECONDARY OUTCOMES:
Study of global survival and progression-free survival according to the results of baseline F-choline PET . | 24 weeks
Study of global survival and progression-free survival at 12 weeks of treatment according to the results of 6 weeks treatment F-choline PET. | 12 weeks
Comparison of Area Under the Curve receiver operating characteristic curve for maximum standardized uptake value (SUVmax) different values. | 12 and 24 weeks
Study of global survival and progression-free survival at 24 weeks of treatment according to the results of 6 weeks treatment F-choline PET. | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe Vuillez, MD PHD, Principal Investigator — University Hospital, Grenoble
Locations (3):
- France (3):
  - Clinique Universitaire d'Oncologie Médicale, CHU de Grenoble, Grenoble
  - Clinique Universitaire de Médecine Nucléaire, CHU de Grenoble, Grenoble
  - Service d'Oncologie Médicale, Institut Daniel Hollard, Groupement Hospitalier Mutualiste, Grenoble

REFERENCES:
- [Background] Jemal A, Siegel R, Ward E, Hao Y, Xu J, Murray T, Thun MJ. Cancer statistics, 2008. CA Cancer J Clin. 2008 Mar-Apr;58(2):71-96. doi: 10.3322/CA.2007.0010. Epub 2008 Feb 20. PMID 18287387
- [Background] Townsend DW. Dual-modality imaging: combining anatomy and function. J Nucl Med. 2008 Jun;49(6):938-55. doi: 10.2967/jnumed.108.051276. Epub 2008 May 15. PMID 18483101
- [Background] Jadvar H. Prostate cancer: PET with 18F-FDG, 18F- or 11C-acetate, and 18F- or 11C-choline. J Nucl Med. 2011 Jan;52(1):81-9. doi: 10.2967/jnumed.110.077941. Epub 2010 Dec 13. PMID 21149473
- [Background] de Jong IJ, Pruim J, Elsinga PH, Vaalburg W, Mensink HJ. 11C-choline positron emission tomography for the evaluation after treatment of localized prostate cancer. Eur Urol. 2003 Jul;44(1):32-8; discussion 38-9. doi: 10.1016/s0302-2838(03)00207-0. PMID 12814672
- [Background] Scattoni V, Picchio M, Suardi N, Messa C, Freschi M, Roscigno M, Da Pozzo L, Bocciardi A, Rigatti P, Fazio F. Detection of lymph-node metastases with integrated [11C]choline PET/CT in patients with PSA failure after radical retropubic prostatectomy: results confirmed by open pelvic-retroperitoneal lymphadenectomy. Eur Urol. 2007 Aug;52(2):423-9. doi: 10.1016/j.eururo.2007.03.032. Epub 2007 Mar 20. PMID 17397992
- [Background] Rinnab L, Mottaghy FM, Blumstein NM, Reske SN, Hautmann RE, Hohl K, Moller P, Wiegel T, Kuefer R, Gschwend JE. Evaluation of [11C]-choline positron-emission/computed tomography in patients with increasing prostate-specific antigen levels after primary treatment for prostate cancer. BJU Int. 2007 Oct;100(4):786-93. doi: 10.1111/j.1464-410X.2007.07083.x. PMID 17822459
- [Background] Giovacchini G, Picchio M, Coradeschi E, Bettinardi V, Gianolli L, Scattoni V, Cozzarini C, Di Muzio N, Rigatti P, Fazio F, Messa C. Predictive factors of [(11)C]choline PET/CT in patients with biochemical failure after radical prostatectomy. Eur J Nucl Med Mol Imaging. 2010 Feb;37(2):301-9. doi: 10.1007/s00259-009-1253-3. Epub 2009 Sep 15. PMID 19756592
- [Background] Giovacchini G, Picchio M, Briganti A, Cozzarini C, Scattoni V, Salonia A, Landoni C, Gianolli L, Di Muzio N, Rigatti P, Montorsi F, Messa C. [11C]choline positron emission tomography/computerized tomography to restage prostate cancer cases with biochemical failure after radical prostatectomy and no disease evidence on conventional imaging. J Urol. 2010 Sep;184(3):938-43. doi: 10.1016/j.juro.2010.04.084. PMID 20643445
- [Background] Breeuwsma AJ, Pruim J, van den Bergh AC, Leliveld AM, Nijman RJ, Dierckx RA, de Jong IJ. Detection of local, regional, and distant recurrence in patients with psa relapse after external-beam radiotherapy using (11)C-choline positron emission tomography. Int J Radiat Oncol Biol Phys. 2010 May 1;77(1):160-4. doi: 10.1016/j.ijrobp.2009.04.090. Epub 2009 Sep 23. PMID 19783375
- [Background] Heinisch M, Dirisamer A, Loidl W, Stoiber F, Gruy B, Haim S, Langsteger W. Positron emission tomography/computed tomography with F-18-fluorocholine for restaging of prostate cancer patients: meaningful at PSA < 5 ng/ml? Mol Imaging Biol. 2006 Jan-Feb;8(1):43-8. doi: 10.1007/s11307-005-0023-2. PMID 16315004
- [Background] Bolla M, de Reijke TM, Van Tienhoven G, Van den Bergh AC, Oddens J, Poortmans PM, Gez E, Kil P, Akdas A, Soete G, Kariakine O, van der Steen-Banasik EM, Musat E, Pierart M, Mauer ME, Collette L; EORTC Radiation Oncology Group and Genito-Urinary Tract Cancer Group. Duration of androgen suppression in the treatment of prostate cancer. N Engl J Med. 2009 Jun 11;360(24):2516-27. doi: 10.1056/NEJMoa0810095. PMID 19516032
- [Background] Bolla M, Collette L, Blank L, Warde P, Dubois JB, Mirimanoff RO, Storme G, Bernier J, Kuten A, Sternberg C, Mattelaer J, Lopez Torecilla J, Pfeffer JR, Lino Cutajar C, Zurlo A, Pierart M. Long-term results with immediate androgen suppression and external irradiation in patients with locally advanced prostate cancer (an EORTC study): a phase III randomised trial. Lancet. 2002 Jul 13;360(9327):103-6. doi: 10.1016/s0140-6736(02)09408-4. PMID 12126818
- [Background] Messing EM, Manola J, Yao J, Kiernan M, Crawford D, Wilding G, di'SantAgnese PA, Trump D; Eastern Cooperative Oncology Group study EST 3886. Immediate versus deferred androgen deprivation treatment in patients with node-positive prostate cancer after radical prostatectomy and pelvic lymphadenectomy. Lancet Oncol. 2006 Jun;7(6):472-9. doi: 10.1016/S1470-2045(06)70700-8. PMID 16750497
- [Background] Tannock IF, de Wit R, Berry WR, Horti J, Pluzanska A, Chi KN, Oudard S, Theodore C, James ND, Turesson I, Rosenthal MA, Eisenberger MA; TAX 327 Investigators. Docetaxel plus prednisone or mitoxantrone plus prednisone for advanced prostate cancer. N Engl J Med. 2004 Oct 7;351(15):1502-12. doi: 10.1056/NEJMoa040720. PMID 15470213
- [Background] Petrylak DP, Tangen CM, Hussain MH, Lara PN Jr, Jones JA, Taplin ME, Burch PA, Berry D, Moinpour C, Kohli M, Benson MC, Small EJ, Raghavan D, Crawford ED. Docetaxel and estramustine compared with mitoxantrone and prednisone for advanced refractory prostate cancer. N Engl J Med. 2004 Oct 7;351(15):1513-20. doi: 10.1056/NEJMoa041318. PMID 15470214
- [Background] de Bono JS, Logothetis CJ, Molina A, Fizazi K, North S, Chu L, Chi KN, Jones RJ, Goodman OB Jr, Saad F, Staffurth JN, Mainwaring P, Harland S, Flaig TW, Hutson TE, Cheng T, Patterson H, Hainsworth JD, Ryan CJ, Sternberg CN, Ellard SL, Flechon A, Saleh M, Scholz M, Efstathiou E, Zivi A, Bianchini D, Loriot Y, Chieffo N, Kheoh T, Haqq CM, Scher HI; COU-AA-301 Investigators. Abiraterone and increased survival in metastatic prostate cancer. N Engl J Med. 2011 May 26;364(21):1995-2005. doi: 10.1056/NEJMoa1014618. PMID 21612468
- [Background] Ryan CJ, Smith MR, de Bono JS, Molina A, Logothetis CJ, de Souza P, Fizazi K, Mainwaring P, Piulats JM, Ng S, Carles J, Mulders PF, Basch E, Small EJ, Saad F, Schrijvers D, Van Poppel H, Mukherjee SD, Suttmann H, Gerritsen WR, Flaig TW, George DJ, Yu EY, Efstathiou E, Pantuck A, Winquist E, Higano CS, Taplin ME, Park Y, Kheoh T, Griffin T, Scher HI, Rathkopf DE; COU-AA-302 Investigators. Abiraterone in metastatic prostate cancer without previous chemotherapy. N Engl J Med. 2013 Jan 10;368(2):138-48. doi: 10.1056/NEJMoa1209096. Epub 2012 Dec 10. PMID 23228172
- [Background] Scher HI, Halabi S, Tannock I, Morris M, Sternberg CN, Carducci MA, Eisenberger MA, Higano C, Bubley GJ, Dreicer R, Petrylak D, Kantoff P, Basch E, Kelly WK, Figg WD, Small EJ, Beer TM, Wilding G, Martin A, Hussain M; Prostate Cancer Clinical Trials Working Group. Design and end points of clinical trials for patients with progressive prostate cancer and castrate levels of testosterone: recommendations of the Prostate Cancer Clinical Trials Working Group. J Clin Oncol. 2008 Mar 1;26(7):1148-59. doi: 10.1200/JCO.2007.12.4487. PMID 18309951
- [Background] Scher HI, Morris MJ, Basch E, Heller G. End points and outcomes in castration-resistant prostate cancer: from clinical trials to clinical practice. J Clin Oncol. 2011 Sep 20;29(27):3695-704. doi: 10.1200/JCO.2011.35.8648. Epub 2011 Aug 22. PMID 21859988
- [Background] Colloca G. Prostate-specific antigen kinetics as a surrogate endpoint in clinical trials of metastatic castration-resistant prostate cancer: a review. Cancer Treat Rev. 2012 Dec;38(8):1020-6. doi: 10.1016/j.ctrv.2012.03.008. Epub 2012 Apr 12. PMID 22503300
- [Background] Effert PJ, Bares R, Handt S, Wolff JM, Bull U, Jakse G. Metabolic imaging of untreated prostate cancer by positron emission tomography with 18fluorine-labeled deoxyglucose. J Urol. 1996 Mar;155(3):994-8. PMID 8583625
- [Background] Fuccio C, Castellucci P, Schiavina R, Guidalotti PL, Gavaruzzi G, Montini GC, Nanni C, Marzola MC, Rubello D, Fanti S. Role of 11C-choline PET/CT in the re-staging of prostate cancer patients with biochemical relapse and negative results at bone scintigraphy. Eur J Radiol. 2012 Aug;81(8):e893-6. doi: 10.1016/j.ejrad.2012.04.027. Epub 2012 May 22. PMID 22621862
- [Background] Beheshti M, Vali R, Waldenberger P, Fitz F, Nader M, Loidl W, Broinger G, Stoiber F, Foglman I, Langsteger W. Detection of bone metastases in patients with prostate cancer by 18F fluorocholine and 18F fluoride PET-CT: a comparative study. Eur J Nucl Med Mol Imaging. 2008 Oct;35(10):1766-74. doi: 10.1007/s00259-008-0788-z. Epub 2008 May 9. PMID 18465129
- [Background] Fuccio C, Schiavina R, Castellucci P, Rubello D, Martorana G, Celli M, Malizia C, Profitos MB, Marzola MC, Pettinato V, Fanti S. Androgen deprivation therapy influences the uptake of 11C-choline in patients with recurrent prostate cancer: the preliminary results of a sequential PET/CT study. Eur J Nucl Med Mol Imaging. 2011 Nov;38(11):1985-9. doi: 10.1007/s00259-011-1867-0. Epub 2011 Jul 6. PMID 21732105
- [Background] Guide pour la rédaction de protocoles pour la tomographie par émission de positons (TEP) à la [18F]-Fluorocholine ([18F]-FCH). Médecine Nucléaire. 2012;36(6):353-9.
- [Background] IRSN. Doses délivrées au patient en scannographie et en radiologie conventionelle - Résultats d'une enquête multicentrique en secteur public. Rapport DRPH/SER N°2010-12. 2010.
- [Background] Daut RL, Cleeland CS, Flanery RC. Development of the Wisconsin Brief Pain Questionnaire to assess pain in cancer and other diseases. Pain. 1983 Oct;17(2):197-210. doi: 10.1016/0304-3959(83)90143-4. PMID 6646795